CLINICAL TRIAL: NCT07140341
Title: A Multi-center, Open Label, Single Arm, Interventional Clinical Study to Assess the Efficacy of ENO Lime in Patients With Ajeerna Vyadhi (Acidity, Acid Indigestion, Indigestion, and Associated Nausea)
Brief Title: A Clinical Study to Assess the Effectiveness of ENO Lime in Participants With Ajeerna Vyadhi (Acidity, Acid Indigestion, Indigestion, and Associated Nausea)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300269
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Indigestion Acid; Indigestion; Nausea
MeSH Terms: conditions — Dyspepsia; Nausea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENO Lime (Experimental): Participants will be instructed to take 1 sachet of ENO Lime powder with approximately 150 milliliters (ml) of normal water as a single dose. Participants will be advised to repeat the dose after 2-hours, if necessary (Maximum 2 sachet per 24-hours). Participants will be followed up for 24-hours.
  Interventions: Drug: ENO Lime

INTERVENTIONS:
Drug: ENO Lime — A fruit salt (sachet of 5-gram powder) with lime flavor containing Svarjiksara (Shudh) 2220 milligram (mg) and Nimbu Rasa (Citrus limon, Fruit Juice Powder) 150 mg

SUMMARY:
The primary purpose of this study is to assess the efficacy of ENO Lime (fruit salt) in participants with Ajeerna vyadhi (acidity, acid indigestion, indigestion, and associated nausea) at 15-minutes after administration of dose. 'Ajeerna vyadhi' is defined as a state of incomplete digestion and metabolism caused due to deranged action of Jatharagni (digestive fire), which leads to the formation of an unprocessed or under-processed state of ingested food termed as Ajeerna.

DETAILED DESCRIPTION:
This will be an open label, single arm, interventional clinical study to evaluate the efficacy and safety of ENO Lime in adult participants with Ajeerna vyadhi (acidity, acid indigestion, indigestion, and associated nausea). The study will be conducted at three sites in India and approximately 40 participants will be enrolled. At baseline, the participants will record the severity of symptoms of Ajeerna vyadhi using the visual analogue scale (VAS) scoring before administering the ENO Lime. As per recommendation, the participants will consume the dose of the ENO Lime on-site and will record any changes in the severity of symptoms of Ajeerna vyadhi using VAS scoring at 2-minutes, 15-minutes, 1-hour, 2-hour post-dose. Participants will be permitted to take the second dose of the ENO Lime (only if required) after 2 hours of the first dose. In such cases, participants will be instructed to record symptoms of Ajeerna vyadhi again using the VAS scoring before taking the second dose (at 0 minutes) and then at 2-minutes, 15-minutes, 1-hour, and 2-hours post-second dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with age 18-60 years (both inclusive).
* Participants newly experiencing symptom/s of Ajeerna vyadhi for not more than 10 days.
* Participants with at least one symptom of Ajeerna vyadhi (according to Charak Samhita and Madhav Nidan) that is acidity (heartburn), acid indigestion (epigastric pain), indigestion (abdominal discomfort), or associated nausea.
* Participants with VAS score greater than or equal to (>=) 40-mm and less than or equal to (<=) 80-mm Ajeerna vyadhi (acidity, acid indigestion, indigestion, or associated nausea) at the Baseline visit.
* Participants are able to read, understand, and provide written informed consent.
* Participants who can understand and complete the VAS.

Exclusion Criteria:

* Participants with chronic and recurrent cases of Ajeerna vyadhi.
* Participants with Updrava of Ajeerna vyadhi (Complications of indigestion).
* Pregnant women (self-reported) and breastfeeding females or females intending to become pregnant during the study.
* Participant had surgery in the last 14 days.
* Participant has been exposed to barium meal 3 days before screening.
* Participants already on any indigestion or acidity medication.
* Participants taking any medicinal/over-the-counter (OTC)/ herbal medicine from the past 3 days.
* Participants on medications that could interact with ENO Lime (example, antacids, proton pump inhibitors, or H2 blockers) as per the judgment of the Investigator/designee.
* Participants with known hypersensitivity to any of the components of ENO Lime (Svarjiksara [Shudh], Nimbu Rasa [Citrus limon, Fruit Juice Powder]).
* Participants with a history of gastrointestinal (GI) disorders such as peptic ulcers, gastritis, irritable bowel syndrome (IBS), or other serious GI diseases.
* Participants with serious renal, hepatic, or cardiovascular diseases.
* Participants on a sodium restricted diet example, those suffering from hypertension or congestive heart failure.
* Participants who have participated in another clinical trial within the last 30 days.
* Any participant who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-09-06 (Actual); Study Completion 2025-09-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Ajeerna Vyadhi (Acidity, Acid Indigestion, Indigestion, And Associated Nausea) Symptoms Using VAS Scoring After 15 Minutes of Taking ENO Lime | Baseline (0-minutes pre-dose) and 15-minutes post-dose on Day 1
  The severity of symptoms of Ajeerna vyadhi will be recorded using VAS scoring. Participants will record a score with a mark at one point along the length of a 100-millimeter (mm) line, where the lowest score 0-mm indicates 'no discomfort' and highest score 100-mm indicates 'worst possible discomfort'. Higher the score, more severe will be the symptoms. Change from baseline will be calculated by subtracting baseline value from the value at 15-minutes.

SECONDARY OUTCOMES:
Change from Baseline in Ajeerna Vyadhi (Acidity, Acid Indigestion, Indigestion, And Associated Nausea) Symptoms Using VAS Scoring After 2-Minutes, 1-Hour, and 2-Hours of Taking ENO Lime | Baseline (0 minutes pre-dose) and 2-minutes, 1-hour, 2-hours post-dose on Day 1
  The severity of symptoms of Ajeerna vyadhi will be recorded using VAS scoring. Participants will record a score with a mark at one point along the length of a 100-mm line, where the lowest score 0-mm indicates 'no discomfort' and highest score 100-mm indicates 'worst possible discomfort'. Higher the score, more severe will be the symptoms. Change from baseline will be calculated by subtracting baseline value from the values at the indicated timepoints.

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Lifepoint Hospital, Pune, Maharashtra
  - Ojas Hospital, Pune, Maharashtra
  - Shri Krishna Super Speciality Institute of Ayurveda, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.